CLINICAL TRIAL: NCT06808893
Title: The Effects of Documentary and Psychiatric Interviewing Methods on Empathy, Attitude and Implicit Association in Psychiatric Nursing Education: A Randomized Controlled Study
Brief Title: The Effects of Documentary and Psychiatric Interviewing Methods in Psychiatric Nursing Education
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 28-01-2025-SK
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Mental Disorder; Stigma of Mental Illness; Nursing Education; Implicit Association Test
Keywords: Baccalaureate Nursing Education; Documentaries and Factual Films; Implicit Bias; Nursing Students; Mentally Ill
MeSH Terms: conditions — Mental Disorders; Bias, Implicit

STUDY DESIGN:
Intervention Model Description: The psychiatric interview group, which is the control group, will have at least one psychiatric interview and will be evaluated with the counselling nurse. The experimental group will have at least one psychiatric interview and the documentary 'Us, You, Them' with patient narratives will be evaluated with a counselling nurse.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (psychiatric interview) (Active Comparator): Nursing students who interview psychiatric patients will be provided with an "Interaction Form" to systematically evaluate and record their interviews. The form is designed to help students analyze their communication processes and document their clinical practice. Before the clinical practice, training on the use of the form will be provided and the points that students should pay attention to in the interviews will be explained. This form consists of the following columns: date and duration of the interview, purpose of the interview, verbal/non-verbal statements of the nurse and patient, effective communication technique and evaluation. During the 6-week psychiatric service practice, students are expected to conduct three psychiatric interviews. After the interviews, students will document the process in detail and will be evaluated by the mentor nurses. Guiding nurses will give feedback to the students, indicating their strengths and areas to improve, and guidance will be provid
  Interventions: Other: Psychiatric interview
- Experimental group (psychiatric interview and documentary) (Experimental): The experimental group was expected to conduct three psychiatric interviews and watch the documentary "Biz,Siz,Onlar" during the 6-week psychiatric service practice. Psychiatric interviews will be carried out with the "Interaction Form" consisting of interview date and duration, purpose of the interview, verbal/nonverbal expressions of the nurse and the patient, effective communication technique and evaluation columns. In addition, students will be shown the documentary "Biz,Siz,Onlar" prepared by the Federation of Schizophrenia Associations of Turkey, which deals with the life stories of schizophrenia patients. The guide nurse will inform the students about the content of the documentary and the viewing process, and students will be encouraged to take notes during the viewing. The documentary, which lasts 56 minutes, will be watched in a quiet environment and then an interactive discussion session will be organized on the themes in the documentary on the clinical practice day.
  Interventions: Other: Psychiatric interview and documentary

INTERVENTIONS:
Other: Psychiatric interview and documentary — Nursing students who interview psychiatric patients will be provided with an "Interaction Form" to systematically evaluate and record their interviews. This form consists of the following columns: date of interview, duration of interview, duration of interview, verbal/non-verbal statements of the nurse and patient, effective communication technique and evaluation. The duration of the interview is expected to be between 30 and 45 minutes. Another component of the combination is the documentary "Us, You, Them" prepared by the Federation of Schizophrenia Associations of Turkey, which deals with the life stories of schizophrenia patients and lasts approximately 56 minutes.
  Arms: Experimental group (psychiatric interview and documentary)
Other: Psychiatric interview — Nursing students who interview psychiatric patients will be provided with an "Interaction Form" to systematically evaluate and record their interviews. This form consists of the following columns: date of interview, duration of interview, duration of interview, verbal/non-verbal statements of the nurse and patient, effective communication technique and evaluation. The duration of the interview is expected to be between 30 and 45 minutes.
  Arms: Control group (psychiatric interview)

SUMMARY:
Negative attitudes towards mental illnesses are an important problem that negatively affects both the social lives of individuals and the effectiveness of health services. Addressing these prejudices, developing empathy and promoting a patient-centred care approach are key goals that can be achieved through clinical experiences and structured educational programmes for nursing students. This single-centre, single-blind, randomised controlled trial aims to examine the effects of documentaries and psychiatric interviews on nursing students' implicit associations, discriminatory attitudes and empathy skills towards mental illnesses. Within the scope of the study, nursing students working in a psychiatric ward will be divided into two groups: one group will work with documentaries including psychiatric interviews and patient narratives, while the other group will only conduct psychiatric interviews. The Implicit Association Test (IAT) and the Attitudes Towards Mental Patients Scale will be used to assess students' implicit associations and attitudes towards psychiatric patients, and the Jefferson Empathy Scale will assess their level of empathy. Data analysis will be performed using SPSS 25.0 software. Given the widespread stigmatisation of psychiatric patients, this study is expected to make a significant contribution to improving the quality of care provided by nursing students in psychiatric settings.

DETAILED DESCRIPTION:
Discrimination and stigmatization towards psychiatric patients remain significant challenges, negatively impacting both individuals' quality of life and their access to healthcare services. These attitudes are not limited to the general public but are also observed among healthcare professionals, including nursing students. Such biases can affect the quality of care provided to psychiatric patients, as nursing students often perceive these individuals as aggressive or dangerous, leading to fear and hesitation in interacting with them. However, studies have shown that clinical placements and mental health education programs can reduce these negative attitudes by fostering empathy and understanding, supporting the development of a patient-centered care approach.

Psychiatric interviews and patient-centered documentaries are effective educational tools to address stigmatization and enhance empathy. Psychiatric interviews provide nursing students with structured opportunities to understand patients' biopsychosocial history, mental health needs, and coping strategies, fostering therapeutic communication skills. Similarly, documentaries featuring personal narratives of psychiatric patients help challenge stereotypes, promote empathy, and deepen students' understanding of mental illnesses. Research shows that combining such methods with academic content, concept mapping, and short films can significantly reduce stigmatization, improve social attitudes, and encourage inclusive practices in healthcare.

This study investigates how psychiatric nursing students' prejudices, discriminatory attitudes, and empathy skills towards mental illnesses can be improved through the use of psychiatric interviews and documentaries. By integrating these innovative approaches into nursing education, the study aims to reduce stigmatization, enhance empathy, and equip future healthcare professionals with the skills necessary to provide inclusive, high-quality care to psychiatric patients. This initiative ultimately seeks to contribute to the long-term improvement of mental health services and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

(1) being a third-year undergraduate student; (2) doing clinical practice in an adult inpatient psychiatric ward; (3) showing normal cognitive functions; (4) having the ability to make sense of visual materials

Exclusion Criteria:

(1) being in clinical practice in community mental health centers and addiction treatment centers; (2) being in clinical practice in special education institutions; (3) having 80% or more absenteeism from clinical practice in adult inpatient psychiatric ward; (4) having 75% or more absenteeism from mental health and psychiatric nursing course; (5) having a psychiatric diagnosis and receiving active treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-02-02 (Estimated)

PRIMARY OUTCOMES:
The Implicit Association Test (IAT) | Within 24 hours after 3 psychiatric interviews and documentary for the experimental group and after 3 psychiatric interviews for the control group
  The Implicit Association Test (IAT), part of Harvard University's Project Implicit, is designed to measure whether psychiatric patients are perceived as dangerous. This test aims to reveal associations that individuals have at an automatic and unconscious level that they do not consciously express. This test, which is especially used for stigmatization studies related to mental health, implicitly measures how dangerous or harmless the participants find psychiatric patients. It examines how quickly participants mentally associate psychiatric patients with positive or negative concepts such as danger or trust. The concepts that are matched faster reflect the implicit attitudes of the person, revealing their unconscious perceptions towards individuals with mental illness.
The Attitudes Towards Mental Patients Scale | Within 24 hours after 3 psychiatric interviews and documentary for the experimental group and after 3 psychiatric interviews for the control group
  The Attitude Towards Mental Patients Scale, developed by Sedat Işıklı in 1998, was prepared to measure a specific psychological construct. The scale consists of 22 items and includes two factors: 'short-term relationships' and 'long-term relationships'. The short-term relationship factors include items 2, 6, 7, 8, 9, 15, 17, 18, 20, 21, and 22. These items reflect attitudes towards shorter-term social relationships in general and towards situations that do not threaten the respondent's personal space. The Long-Term Relationships Factor includes items 1, 3, 4, 5, 10, 11, 12, 13, 14, 16, and 19 and assesses attitudes towards longer-term and closer relationships. The scale is scored on a 5-point Likert scale: 5=Strongly agree, 4=Agree, 3=No opinion, 2=Disagree, and 1=Strongly disagree. High scores indicate a positive attitude.

SECONDARY OUTCOMES:
Jefferson Empathy Scale | Within 24 hours after 3 psychiatric interviews and documentary for the experimental group and after 3 psychiatric interviews for the control group
  The original form of the scale was developed by Hojat et al. in 2001 to measure the empathy level of health professionals in patient care. The adaptation study of the scale into Turkish was conducted by Yanık and Saygılı in 2014. The scale, which consists of a total of 20 items and three sub-dimensions, is a 7-point Likert type. Participants rate the level of empathy between 1 (strongly disagree) and 7 (strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bilge A, Palabiyik O. The Effect of Short Films About Mental Health and Disorders on Preventing Stigmatization in Nursing Education. Arch Psychiatr Nurs. 2017 Feb;31(1):88-92. doi: 10.1016/j.apnu.2016.09.006. Epub 2016 Sep 8. PMID 28104066
- [Result] Li, Y., 2016. From "whom to blame" to "nothing to fear": documentary narratives, voices, and "dependent destigmatization" of severe mental patients (SMPs) in Hong Kong. Chin. J. Commun. 9 (4), 403-421. https://doi.org/10.1080/17544750.2016.1202293.
- [Result] Yildiz E. What Do Nursing Students Tell Us About Their Communication With People With Mental Illness? A Qualitative Study. J Am Psychiatr Nurses Assoc. 2021 Nov-Dec;27(6):471-482. doi: 10.1177/1078390319892311. Epub 2019 Dec 3. PMID 31795795
- [Result] Chou HJ, Tseng KY. The Experience of Emergency Nurses Caring for Patients with Mental Illness: A Qualitative Study. Int J Environ Res Public Health. 2020 Nov 18;17(22):8540. doi: 10.3390/ijerph17228540. PMID 33217909
- [Result] Todorova L, Johansson A, Ivarsson B. Perceptions of ambulance nurses on their knowledge and competence when assessing psychiatric mental illness. Nurs Open. 2021 Mar;8(2):946-956. doi: 10.1002/nop2.703. Epub 2020 Nov 27. PMID 33570281
- [Result] Ciydem E, Avci D. Effects of the psychiatric nursing course on students' beliefs toward mental illness and psychiatric nursing perceptions in Turkey. Perspect Psychiatr Care. 2022 Jan;58(1):348-354. doi: 10.1111/ppc.12796. Epub 2021 Apr 8. PMID 33834489
- [Result] Happell B, Gaskin CJ. The attitudes of undergraduate nursing students towards mental health nursing: a systematic review. J Clin Nurs. 2013 Jan;22(1-2):148-58. doi: 10.1111/jocn.12022. Epub 2012 Nov 21. PMID 23170825
- [Result] Sideras, S., McKenzie, G., Noone, J., Dieckmann, N.F., Allen, T.L., 2015. Impact of a simulation on nursing students' attitudes toward schizophrenia. Clin. Simul. Nurs. 11 (2), 134-141. https://doi.org/10.1016/j.ecns.2014.11.005.
- [Result] Šimičić, M., 2023. Nurses' attitudes and stigma about mental illness and substance abuse. Open Access Maced. J. Med. Sci. 11 (G), 98-104. https://doi.org/10.3889/oamjms.2023.11713.
- [Result] Porfyri GN, Athanasiadou M, Siokas V, Giannoglou S, Skarpari S, Kikis M, Myroforidou A, Anoixa M, Zerakis N, Bonti E, Konsta A, Diakogiannis I, Rudolf J, Deretzi G. Mental health-related stigma discrimination and prejudices among Greek healthcare professionals. Front Psychiatry. 2022 Nov 30;13:1027304. doi: 10.3389/fpsyt.2022.1027304. eCollection 2022. PMID 36532175
- [Result] Kohn L, Christiaens W, Detraux J, De Lepeleire J, De Hert M, Gillain B, Delaunoit B, Savoye I, Mistiaen P, Jespers V. Barriers to Somatic Health Care for Persons With Severe Mental Illness in Belgium: A Qualitative Study of Patients' and Healthcare Professionals' Perspectives. Front Psychiatry. 2022 Jan 26;12:798530. doi: 10.3389/fpsyt.2021.798530. eCollection 2021. PMID 35153863
- [Result] Diatmika, I.P., Karmila, D., 2022. Stigma influence of the outcome (experiences, motivations, and obstacles) towards people with mental illness problems in Babaka Public Health Centre, Lombok. Berk. Kedokteran 18 (2), 161. https://doi.org/10.20527/jbk.v18i2.14492.
- [Result] Zhang Z, Sun K, Jatchavala C, Koh J, Chia Y, Bose J, Li Z, Tan W, Wang S, Chu W, Wang J, Tran B, Ho R. Overview of Stigma against Psychiatric Illnesses and Advancements of Anti-Stigma Activities in Six Asian Societies. Int J Environ Res Public Health. 2019 Dec 31;17(1):280. doi: 10.3390/ijerph17010280. PMID 31906068
- [Result] Singh GP, Chavan BS, Kaur P, Bhatia S. Physical illnesses among psychiatric outpatients in a tertiary care health institution: A prospective study. Indian J Psychiatry. 2006 Jan;48(1):52-5. doi: 10.4103/0019-5545.31620. PMID 20703416
- [Result] Rymaszewska J, Jarosz-Nowak J, Kiejna A, Kallert T, Schutzwohl M, Priebe S, Wright D, Nawka P, Raboch J. Social disability in different mental disorders. Eur Psychiatry. 2007 Apr;22(3):160-6. doi: 10.1016/j.eurpsy.2006.11.006. Epub 2007 Jan 16. PMID 17227704
- [Result] Angermeyer MC, van der Auwera S, Carta MG, Schomerus G. Public attitudes towards psychiatry and psychiatric treatment at the beginning of the 21st century: a systematic review and meta-analysis of population surveys. World Psychiatry. 2017 Feb;16(1):50-61. doi: 10.1002/wps.20383. PMID 28127931
- [Derived] Koroglu Gokbel S, Durat G. The Effects of Documentary and Psychiatric Interviewing Methods on Empathy, Attitude, and Implicit Association in Psychiatric Nursing Education: A Randomized Controlled Study. West J Nurs Res. 2026 Feb;48(2):162-174. doi: 10.1177/01939459251392988. Epub 2025 Dec 17. PMID 41404938